CLINICAL TRIAL: NCT04741217
Title: A Proof of Concept Study to Evaluate Aerosol Generation During Non-Invasive Positive Pressure Respiratory Procedures
Brief Title: Aerosolisation During Respiratory Procedures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 288629
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2020-08

CONDITIONS: Healthy; Respiratory Tract Infections; Lung Infection; Droplet Spread
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not an interventional study — No interventions are implemented. This is an observational study of respiratory droplet aerosolisation during respiratory procedures.

SUMMARY:
Currently, a major issue within respiratory medicine is undertaking procedures that generate aerosolisation with the concern of spreading infection, such as the SARS-COV-2/COVID-19 virus. It is anecdotally reported that lung function testing and positive airways pressure devices used in clinical practice are aerosol generating procedures however the data to support this is limited. With the advent of high-speed imaging systems that can capture and quantify particle size and velocity we aim to investigate the aerosol generation in routine non-invasive positive pressure respiratory procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Healthy subjects with no active medical conditions or previous pneumothorax
* Cognitively and linguistically able to follow instructions given in English and provide informed consent

Exclusion Criteria:

* Significant respiratory, cardiac or neurological conditions or previous pneumothorax
* Smoking history greater than 10 pack years
* Acute illness at the time of assessment
* Allergies to latex, metals or local anaesthetic agents

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Characterisation of aerosolised respiratory droplets | 1 year
  Performed using high-speed imaging and particle size counters

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be shared based upon consideration of reasonable requests from researchers with a stated objective.